CLINICAL TRIAL: NCT00046826
Title: A Phase II Clinical Trial of Taxotere, Emcyt and Thalidomide (TET) for the Treatment of Hormone-Refractory Prostate Cancer
Brief Title: Docetaxel, Estramustine, and Thalidomide in Treating Patients With Prostate Cancer Previously Treated With Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nuvance Health (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069081; NH-0139; NCI-V01-1681
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2006-01

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Estramustine; Thalidomide

INTERVENTIONS:
Drug: docetaxel
Drug: estramustine phosphate sodium
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may stop the growth of prostate cancer by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with thalidomide may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining docetaxel and estramustine with thalidomide in treating patients who have prostate cancer previously treated with hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in patients with hormone-refractory prostate cancer treated with docetaxel, estramustine, and thalidomide.
* Determine the safety and toxicity of this regimen in these patients.
* Determine the efficacy of this regimen for pain control in these patients.

OUTLINE: Patients receive oral estramustine on days 1-3 and docetaxel IV over 1 hour on day 2 for 3 weeks. Treatment repeats every 4 weeks for at least 6 courses in the absence of disease progression or unacceptable toxicity.

Patients also receive oral thalidomide once daily beginning on day 1 and continuing for 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly until disease progression.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Prior treatment with androgen ablation including:

  * Orchiectomy OR
  * Luteinizing hormone-releasing hormone (LHRH) therapy (e.g., leuprolide)

    * Patients on leuprolide must continue to receive the drug
* Prior nonsteroidal antiandrogens (e.g., flutamide, bicalutamide, or nilutamide) required
* Metastatic disease with disease progression during androgen ablation, defined by at least 1 of the following:

  * 2 consecutive increased prostate-specific antigen (PSA) levels measured at least 1 week apart
  * More than 25% increase in bidimensionally measurable soft tissue metastases
  * 20% increase in the sum of the baseline sum of longest diameter of measurable lesions
  * Appearance of new lesions
  * Appearance of new foci on a radionuclide bone scan
* PSA greater than 10 ng/dL
* Testosterone no greater than 50 ng/mL (castrate level)
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 16 weeks

Hematopoietic:

* WBC greater than 3,500/mm3
* Absolute neutrophil count greater than 1,500/mm3
* Platelet count greater than 100,000/mm3
* Hemoglobin at least 8 g/dL

Hepatic:

* AST and/or ALT no greater than 2.5 times upper limit of normal (ULN) if alkaline phosphatase no greater than ULN OR
* Alkaline phosphatase no greater than 4 times ULN if AST/ALT no greater than ULN
* Bilirubin no greater than ULN

Renal:

* Creatinine less than 2.2 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart disease
* No history of arterial or venous thrombosis
* No cerebrovascular accident within the past year

Pulmonary:

* No history of pulmonary embolism

Other:

* Fertile patients must use effective contraception during and for 4 weeks after study
* No peripheral neuropathy grade 2 or greater
* No active infection
* No serious concurrent medical illness that would preclude study
* No prior severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No other prior or concurrent active malignancy within the past 2 years except non-melanoma skin cancers
* No other medical condition or reason that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for prostate cancer

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior flutamide (6 weeks for bicalutamide or nilutamide) and continued evidence of disease progression (rising PSA)
* Prior steroids for prostate cancer allowed
* No concurrent steroids except for pre-medication for docetaxel

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No concurrent herbal supplements to treat prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2007-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate as measured by RECIST criteria and prostate-specific antigen (PSA) response 3 months, 6 months, and 1 year after treatment

SECONDARY OUTCOMES:
Safety and toxicity as measured by CTC toxicity grading at baseline and during every visit
Effectiveness of taxotere, emcyt, and thalidomide in pain control as measured by the pain scale at baseline and during every visit

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Frank, MD, Study Chair — Nuvance Health
Locations (2):
- United States (2):
  - Whittingham Cancer Center at Norwalk Hospital, Norwalk, Connecticut
  - Carl and Dorothy Bennett Cancer Center at Stamford Hospital, Stamford, Connecticut

REFERENCES:
- [Result] Frank RC, Coscia A, Versea L, et al.: Low dose docetaxel, estramustine and thalidomide followed by maintenance thalidomide for the treatment of hormone refractory prostate cancer (HRPC): a phase II community based trial. [Abstract] J Clin Oncol 22 (Suppl 14): A-4681, 426s, 2004.